CLINICAL TRIAL: NCT03046719
Title: Subconjunctiva Bupivacaine as Analgesia in Intravitreal Silicone Oil Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Aida Rosita Tantri SpAn-KA, Consultant, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IndonesiaUAnes009
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Retinal Detachment
Keywords: bupivacaine; intravitreal; analgesia; silicone oil removal; retinal detachment; subconjunctival
MeSH Terms: conditions — Retinal Detachment; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Bupivacaine 0,5% (Active Comparator): Subjects received subconjunctival bupivacaine 0,5% 2,5ml in between stitches.
  Interventions: Drug: Bupivacaine 0,5%
- NaCl 0,9% (Placebo Comparator): Subjects received subconjunctival NaCl 0,9% in between stitches.
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: Bupivacaine 0,5% — Bupivacaine 0,5% was given on the subconjunctiva, in between stitches by the surgeon after finishing the last stitches
  Arms: Bupivacaine 0,5%
Drug: NaCl 0,9% — NaCl 0,9% was given on the subconjunctiva, in between stitches by the surgeon after finishing the last stitches
  Arms: NaCl 0,9%

SUMMARY:
The study aimed to investigate the effectivity of bupivacaine 0,5% as post-operative analgesia in intravitreal silicone evacutaion surgery

DETAILED DESCRIPTION:
Approval from Ethical Committee of Faculty of Medicine Universitas Indonesia was acquired prior conducting the study. Subjects were given informed consent before enrolling the study and randomized into two groups. Intravenous (IV) cannule with Ringer Lactate fluid, non-invasive blood pressure monitor, electrocardiogram (ECG) and pulse-oxymetry were set on the subjects in the operation room. Co-induction was done with midazolam 0,05 mg/kg and fentanyl 2 mcg/kg. Induction was done with propofol 1-2 mg/kg, followed by Laryngeal Mask insertion facilitated by atracurium 0,5 mg/kg. Maintenance was done with sevoflurane 1-2 vol%, O2:H2O = 1:2, flow 2 liter/minute. Surgery started. After final stitching, Group 1 received subconjunctival bupivacaine 0,5% 2,5ml in between stitches; Group 2 received subconjunctival NaCl 0,9% in between stitches. Both groups received paracetamol 20 mg/kgBW IV as post-operative analgesics. Hemodynamic, pain degree (using Visual Analog Scale / VAS), and nausea/vomiting incidence, and the time for first requested additional analgesia were recorded. Data was analyzed using SPSS (Statistical Package for Social Scientist), for numerical data using unpaired T-test or Mann-Whitney-U test, for categorical data using Chi-square test or Fischer Exact's Test. Data normality was tested by Kolmogorov-Smirnov test. Significant value is p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-60 years old, with ASA physical status I-II and BMI 18,5-30 kg/m2 who were planned to do intravitreal silicone evacuation surgery.
* Subjects have been explained about the study, have agreed to enroll and have signed the informed consent form

Exclusion Criteria:

* Subjects with history of post-operative chronic pain
* Subjects with history of pre-operative long term use of analgesic
* Subjects with history of local anesthetics allergy, pregnant subjects
* Subjects with ambulation operation
* Subjects with glaucoma or ocular hypertension
* Subjects with cognition dysfunction or communication disturbance
* Subjects with additional surgery other than silicone oil removal

Drop Out criteria:

* Subjects with intraoperative complications (e.g. shock, anaphylactic reaction, seizures, severe respiratory disturbance)
* Subjects with post-operative intraocular pressure > 22mmHg.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The degree of pain | 2 months
  The degree of pain was measured in the morning after the surgery by Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
The time for first requested post-operative additional analgesia | 2 months
  The time for first requested post-operative additional analgesia was measured in minutes in the morning after the surgery
Side Effects | 2 months
  post-operative nausea / vomiting incidence

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Central National Hospital, Central Jakarta, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Fekrat S, Elsing SH, Raja SC, Campochiaro PA, de Juan E Jr, Haller JA. Eye pain after vitreoretinal surgery: a prospective study of 185 patients. Retina. 2001;21(6):627-32. doi: 10.1097/00006982-200112000-00010. PMID 11756886
- [Background] Bartley EJ, Fillingim RB. Sex differences in pain: a brief review of clinical and experimental findings. Br J Anaesth. 2013 Jul;111(1):52-8. doi: 10.1093/bja/aet127. PMID 23794645
- [Background] Wandner LD, Scipio CD, Hirsh AT, Torres CA, Robinson ME. The perception of pain in others: how gender, race, and age influence pain expectations. J Pain. 2012 Mar;13(3):220-7. doi: 10.1016/j.jpain.2011.10.014. Epub 2012 Jan 5. PMID 22225969
- [Background] Fillingim RB, King CD, Ribeiro-Dasilva MC, Rahim-Williams B, Riley JL 3rd. Sex, gender, and pain: a review of recent clinical and experimental findings. J Pain. 2009 May;10(5):447-85. doi: 10.1016/j.jpain.2008.12.001. PMID 19411059
- [Background] Belmonte C, Aracil A, Acosta MC, Luna C, Gallar J. Nerves and sensations from the eye surface. Ocul Surf. 2004 Oct;2(4):248-53. doi: 10.1016/s1542-0124(12)70112-x. PMID 17216099